CLINICAL TRIAL: NCT02908061
Title: A Prospective, Randomized Trial of Preventive Mesh Placement at the Time of Radical Cystectomy to Reduce the Chances of Developing a Parastomal Hernia
Brief Title: A Study to Determine if Mesh Placement During Bladder Surgery Can Reduce the Chances of Developing a Hernia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1285
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2024-09

CONDITIONS: Radical Cystectomy
Keywords: Mesh Placement; Radical Cystectomy; 16-1285

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Surgery (Usual approach group) (Active Comparator): standard surgery
  Interventions: Procedure: Surgery Radical Cystectomy
- Surgery + Mesh Placement (Experimental): prophylactic mesh at the time of standard surgery
  Interventions: Procedure: Surgery Radical Cystectomy; Procedure: Ultrapro mesh

INTERVENTIONS:
Procedure: Surgery Radical Cystectomy — All surgeries will be performed in an open or laparoscopic fashion.
Procedure: Ultrapro mesh — Surgery Mesh Placement. All surgeries will be performed in an open or laparoscopic fashion.
  Arms: Surgery + Mesh Placement

SUMMARY:
The purpose of this study is to compare any good and bad effects of using Ultrapro mesh along with the usual bladder removal surgery, versus having the usual bladder removal surgery without the use of the mesh.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing RC and IC formation in an elective setting,for cancer.

Exclusion Criteria:

* Expected survival < 12 months
* Salvage RC
* Distant metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of radiographic Parastomal Hernia | within 2 years of RC and IC.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bochner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and follow-up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and follow-up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and follow-up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent only and Follow Up), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/